CLINICAL TRIAL: NCT04161846
Title: Reaching Racial/Ethnic Minority Communities to Support Healthy Lifestyle Change: Virtual World Training for Community Health Workers
Brief Title: Virtual World Training for Community Health Workers (CHW)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Laurie Ruggiero, Ph.D., Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1106606-8
Record Dates: First submitted 2019-06-18; First posted 2019-11-13 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus Risk

STUDY DESIGN:
Intervention Model Description: Randomized 2 group repeated measures design (Pre-Pandemic) [Pandemic modification: Only Virtual world group]
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual World Program (Experimental): Participants take part in a group training delivered using a virtual world approach.
  Interventions: Behavioral: Virtual Training
- In Person Program (Active Comparator): Participants take part in a group training delivered using an in person approach.
  Interventions: Behavioral: In Person Training

INTERVENTIONS:
Behavioral: Virtual Training — The intervention involves a CHW training focused on raising awareness of diabetes prevention in the community. It is delivered remotely over 10 weeks using an internet based approach.
  Arms: Virtual World Program
Behavioral: In Person Training — The intervention involves a CHW training focused on raising awareness of diabetes prevention in the community. It is delivered in person over 10 weeks.
  Arms: In Person Program

SUMMARY:
Standard, effective, and scalable training models are needed to help equip community health workers in their community-based diabetes prevention awareness efforts. This study will tailor/adapt, implement, and evaluate an innovative internet-based virtual world model to remotely deliver a diabetes prevention awareness training program to community health workers.

DETAILED DESCRIPTION:
Standard, effective, and scalable training models are needed to help equip community health workers in their community-based diabetes prevention awareness efforts. This study will tailor/adapt, implement, and evaluate an innovative internet-based virtual world model to remotely deliver a diabetes prevention awareness training program to community health workers. A sequential mixed-methods design is used to address these specific aims: 1. Use community-based participatory research methods to guide the overall study and inform tailoring and adaptation of our virtual world model to deliver the CHW training program; 2. Conduct a randomized pilot study to compare change in primary outcomes (0, 12 weeks) after the in-person versus virtual world delivery of the program; and 3. Conduct summative focus groups to gather information to refine the program and study methodology.

ELIGIBILITY:
Inclusion Criteria:

* community health worker
* 18-65 years old
* Female
* Of African American/Black/African ancestry
* not getting 150 minutes of physical activity weekly and/or overweight
* residing in Chicago/driving distance to Chicago study site
* regular access to internet and computer

Exclusion Criteria:

• does not meet inclusion criteria

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Only
Enrollment: 26 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Change in content knowledge will be measured using the program Knowledge Questionnaire | Following program completion (10-12 weeks)
  Program content knowledge will be assessed using an adapted version of the original training program knowledge questionnaire. Scores represent the number of content questions answered correctly. Higher scores represent greater program knowledge.
Post Training Presentation Delivery Skills | Following program completion (10-12 weeks)
  Each CHW will be asked to prepare and deliver a brief presentation, including 3 standardized topic areas.

SECONDARY OUTCOMES:
Change in Lifestyle Habits | Following program completion (10-12 weeks)
  Eating habits will be assessed using the Visually-Enhanced Food Behavior Checklist.
Change in Physical Activity | Following program completion (10-12 weeks)
  Physical activity will be assessed with International Physical Activity Questionnaire (IPAQ).

OTHER OUTCOMES:
Change in self-efficacy and Stage of Change. A Self-Efficacy Index will be used and Stage of Change individual questions will be used for healthy eating and physical activity. | Following program completion (10-12 weeks)
  A multi-item index of self-efficacy will be used to examine confidence in making lifestyle changes and in delivering the content. Higher scores represent greater confidence. Stage of change questions will assess CHW motivation (i.e., pre-contemplation, contemplation, preparation) or achievement of eating habit and physical activity behaviors (i.e., action/maintenance stages).
Adherence | During training sessions (up to 10 weeks).
  Attendance will be measured by a count of the number of training sessions attended.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Ruggiero, Ph.D, Principal Investigator — University of Delaware
Locations (1):
- UIC College of Nursing, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No